CLINICAL TRIAL: NCT00851279
Title: Stereotaxis Study To Obliterate Persistent Ventricular Tachycardia: Data Collection of Clinical Scar-related VT Cases
Brief Title: Stereotaxis Study To Obliterate Persistent Ventricular Tachycardia
Acronym: STOP-VT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stereotaxis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM-CLIN-013
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-07

CONDITIONS: Ventricular Tachycardia
Keywords: arrhythmia; ventricular tachycardia; ablation; mapping; electrophysiology
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic irrigated ablation catheter (Experimental): Patients with documented VT and prior MI, in whom an ICD was implanted either for primary or secondary prevention, were recruited for endocardial mapping/ablation during VT (entrainment mapping, activation mapping) and/or substrate mapping in sinus rhythm (elimination of fractionated/late potentials, endocardial scar homogenization) with remote magnetic navigation (Niobe, Stereotaxis Inc.,St Louis, USA) and irrigated RF ablation (NaviStar RMT ThermoCool, Biosense Webster,California, USA).
  Interventions: Device: Magnetic irrigated ablation catheter

INTERVENTIONS:
Device: Magnetic irrigated ablation catheter — Magnetic irrigated catheter to be used with the magnetic navigation system
  Other Names: Niobe; Stereotaxis; Navigant

SUMMARY:
This is a prospective, non-randomized, multi-center clinical case series evaluating the outcomes of the magnetic navigation system in ventricular tachycardia (VT) cases. Subjects will be evaluated acutely and will be followed clinically at 1, 6 and 12 months post-treatment.

DETAILED DESCRIPTION:
Catheter ablation of ventricular tachycardia (VT) is greatly facilitated by using a substrate mapping approach - that is, mapping of the left ventricle during sinus or paced rhythm to identify diseased myocardium. Using three dimensional electroanatomical mapping, it is possible to reconstruct an anatomical rendering of the left ventricle based on voltage. For hemodynamically stable or unstable VTs, various electrophysiologic maneuvers can then be used to identify the critical portions of the VT circuit within the scar (entrainment mapping, identification of diastolic potentials, identification of electrically-unexcitable scar, fractionated potentials and pace mapping).

These methods are limited by the resolution of the substrate map, accuracy of catheter manipulation, and operator skill. To this end, a magnetic navigation system has been developed that allows for remote cardiac mapping. When used in concert with a compatible electroanatomical mapping system, it is possible to create a high-density ventricular substrate map of healed myocardial infarction. By removing the necessity for technical skill with catheter manipulation, this system has the potential for both improving the efficacy of VT ablation and expanding the clinical use of this substrate mapping approach.

Recently, a higher-powered, irrigated tip catheter has become available in certain markets for use in cardiac arrhythmia ablations. This study will evaluate the outcomes of using this magnetic irrigation ablation catheter during mapping and ablation of VT while also using remote magnetic navigation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between the ages of 18 - 80 years
* Willing to provide prior written informed consent per local ethics committee guidelines
* Subjects must present with ventricular tachycardia, characterized by: history of myocardial scar and spontaneous ventricular tachycardia
* Able to be safely exposed to static magnetic fields
* No in-situ devices are present or any in-situ devices have been verified to be compatible to magnetic fields

Exclusion Criteria:

* Presence of a mobile ventricular thrombus
* Inability to access the left ventricle
* Subjects must not have any contraindications to short-term anticoagulation
* Subjects must not have a life expectancy of <1 year due to a medical illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, Principal Investigator — Na Homolce Hospital, Prague, CZ
Locations (4):
- United States (2):
  - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Na Homolce Hospital, Prague, Czechia
- Herzzentrum Universitat Leipzig, Leipzig, Germany

REFERENCES:
- See also: Study Sponsor — http://www.stereotaxis.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnetic Irrigated Ablation Catheter: Magnetic irrigated catheter for VT: Magnetic irrigated catheter to be used with the magnetic navigation system
Period: Overall Study
Arm/Group | Magnetic Irrigated Ablation Catheter
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Magnetic Irrigated Ablation Catheter: Patients underwent ablation therapy using remote magnetic navigation, RMN (Niobe, Stereotaxis Inc.,St Louis, USA), and an irrigated RF ablation catheter (NaviStar RMT ThermoCool, Biosense Webster,California, USA).
Arm/Group | Magnetic Irrigated Ablation Catheter
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 33
Age, Continuous [Median (Standard Deviation); unit: years] | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 12
  Czech Republic | 32
  Germany | 9
Left Ventricular Ejection Fraction [Mean (Inter-Quartile Range); unit: percent] | 31.5 [25 to 40]
History of cerebro-vascular accident (CVA) [Number; unit: participants] | 9
History of transient ischemic attack (TIA) [Number; unit: participants] | 3
History of diabetes [Number; unit: participants] | 16
Pre-procedural arrhythmia treatment with beta-blockers [Number; unit: participants] | 47
Pre-procedural arrhythmia treatment with amiodarone [Number; unit: participants] | 34
ICD implanted prior to the ablation procedure [Number; unit: participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free From VT at 1 Year Post-Treatment
Description: In order to qualify for inclusion in the chronic success statistic, patients must first be an acute success and must have had no VTs identified in their ICD history post ablation therapy.
Time Frame: 1 Year follow-up
Measure: Number; unit: percentage of participants free from VT
Groups:
- Magnetic Irrigated Ablation Catheter: Either the transseptal or transaortic approach was employed to gain access for endocardial mapping/ablation during VT (entrainment mapping, activation mapping) and/or substrate mapping in sinus rhythm (elimination of fractionated/late potentials, endocardial scar homogenization) with RMN (Niobe, Stereotaxis Inc.,St Louis, USA) and irrigated RF ablation (NaviStar RMT ThermoCool, Biosense Webster,California, USA).
Arm/Group | Magnetic Irrigated Ablation Catheter
Number analyzed (Participants) | 53
percentage of participants free from VT | 62

ADVERSE EVENTS:
Groups:
- Magnetic Irrigated Ablation Catheter: Magnetic irrigated catheter for VT: Magnetic irrigated catheter to be used with the magnetic navigation system
  There were no adverse events associated with the procedure and within a 7 to 10 days post-doc window
Arm/Group | Magnetic Irrigated Ablation Catheter
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days